CLINICAL TRIAL: NCT02704598
Title: Comparison of the Recanalization Rate and Incidence of Postthrombotic Syndrome in Patients With Lower-limb Deep Venous Thrombosis Treated With Rivaroxaban or Warfarin
Brief Title: Comparison Between Xarelto Versus Warfarin in the Recanalization Rate of Deep Venous Thrombosis in Patients Legs.
Acronym: DVT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital do Servidor Publico Estadual (Other)
Responsible Party: Principal Investigator, Rafael de Athayde Soares, Dr. Rafael de Athayde Soares, MD, Hospital do Servidor Publico Estadual
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2016-02-28; First posted 2016-03-10 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Deep Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Active Comparator): Patients with deep venous thrombosis using Rivaroxaban for 6 months, and then will be evaluated with DUPLEX SCAN to assess the recanalization rate, and also the clinical signs and symptoms.
  Interventions: Drug: Rivaroxaban
- Warfarin (Active Comparator): Patients with deep venous thrombosis using Warfarin for 6 months, and then will be evaluated wiht DUPLEX SCAN to assess the recanalization rate, and also the clinical signs and symptoms.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Evaluate the efficacy of the oral anticoagulants in the treatment of deep venous tromboses, assessing clinical signs and symptoms, as so the recanalization rate using DUPLEX SCAN.
  Other Names: xarelto
  Arms: Rivaroxaban
Drug: Warfarin — Evaluate the efficacy of the oral anticoagulants in the treatment of deep venous tromboses, assessing clinical signs and symptoms, as so the recanalization rate using DUPLEX SCAN.
  Other Names: Marevan
  Arms: Warfarin

SUMMARY:
This is a prospective, randomized study, aiming to evaluate patients with Deep Venous Thrombosis in lower limbs and the recanalization rates evaluated with DUPLEX ultrasound, as so the clinical outcomes in patients submitted to oral anticoagulation with Rivaroxaban versus Warfarin.

DETAILED DESCRIPTION:
This study was approved by the Research Ethics Committee of the Hospital do Servidor Público Estadual, São Paulo, Brazil, and was registered at clinicaltrials.gov under NCT 02704598. This prospective, randomized, consecutive, double-blind cohort study included patients treated for acute iliofemoral and/or femoropopliteal DVT of a lower limb at the Division of Vascular and Endovascular Surgery, Hospital do Servidor Público Estadual, São Paulo, Brazil, between march 2016 and July 2018. The patient data were collected during an appointment at the routine follow-up, and recorded with the proper protocols. The data obtained included the patient's general and demographic characteristics, and the information recorded during the outpatient follow-up visits. This research received no specific funding.

The noninclusion criteria were: pregnancy, age < 18 years or > 80 years, chronic renal failure, chronic hepatic chronic failure, inferior vena cava thrombosis, contraindication for any type of anticoagulation, previous DVT on the ipsilateral affected limb, or any type of active cancer, and patients who refused to participate in the study.

The exclusion criteria were: several hemorrhagic complications that required the discontinuation of anticoagulation, death after < 30 days, allergic reaction to any anticoagulant, a diagnosis of active cancer during follow-up, loss to follow-up, difficulty in achieving proper anticoagulation due to patient nonadherence to the treatment protocol, and incomplete data.

The diagnosis of DVT was made with clinical signs and symptoms, laboratory tests such as D-dimer, and routine DUS of the affected limb. The criteria used to confirm acute DVT with DUS were the absence or diminution of venous flow, incompressibility of the vessel, visible thrombus, enlarged vein diameter, immobility of the valves, and loss of respiratory phasicity.13 All the patients diagnosed with acute DVT were hospitalized and received initial anticoagulation with subcutaneous enoxaparin (1 mg/kg/dose) every 12 h (12/12 h) or intravenous unfractionated heparin (IUH) (loading dose 80 UI/kg, and 18 UI/kg/h) for at least 48-72 h. The infusion dose of IUH was adjusted to achieve the therapeutic activated partial thromboplastin time (APTT) established by the hospital laboratory within every 4-6 h period. After initial admission, the patients were randomized into two groups: group 1 patients received oral rivaroxaban, with a loading dose of 15 mg 12/12 h for 21 days after the initial dose, and 20 mg/day for 6 months; group 2 patients received oral warfarin, sufficient to maintain an INR of 2-3 for 6 months. The patients in group 2 were kept in hospital on subcutaneous enoxaparin or intravenous unfractionated heparin until their INR was 2-3. The patients were discharged after their INR achieved the therapeutic dose.

During the follow-up visits, all the patients were subjected to a DUS analysis by a physician blinded to the type of drug therapy, with defined protocols that assessed the compressibility of the external iliac vein, common femoral vein, superficial femoral vein, and popliteal vein. Flow recanalization was evaluated by confirming the total vein flow, the partial vein flow, or the absence of vein flow. All vessels evaluated were tested for the absence or presence of reflux and the grade of reflux.

The following ultrasound criteria were used to determine absence of recanalization flow: partial compressibility of the vein, diminution of the vessel diameter, heterogeneous and hyperechoic thrombus, multiple channels of flow inside the veins, reflux, and collateral circulation.13 All the patients were followed-up with outpatient visits at 1, 3, 6, and 12 months after discharge. The following information was recorded at each visit: physical examination, DUS and laboratory tests, such as D-dimer, for all patients, and INR for patients receiving warfarin. The patients in group 2 were seen once a week to ensure that their INR remained at 2-3 and to confirm adequate anticoagulation. At the physical examination, the thigh was measured with a tape measure in the medium segment and the legs in the proximal segments, to record their diameters, in order to objectively assess the improvement in the swelling and edema of the leg.

A diagnosis of PTS was made with the Villalta scale when the patient's symptoms had remained unresolved for 6 months after treatment.9 The scale's components (five symptoms and six signs) are each rated on a 4-point severity scale, and the points are summed to produce a total score. A score > 4 indicates PTS. The five symptoms (pain, cramps, heaviness, pruritus, and paresthesia) were assessed by patient self-report, and the six signs (edema, skin induration, hyperpigmentation, venous ectasia, redness, and pain during calf compression) by a clinician. The severity of each symptom and sign was rated as 0 (absent), 1 (mild), 2 (moderate), or 3 (severe). These were summed to yield the total Villalta PTS score: 0-4, no PTS; 5-9, mild PTS; 10-14, moderate PTS; ≥ 15 or presence of an ulcer, severe PTS.

The purpose of this study was to examine the long-term outcomes (after 12 months) in two groups of patients after treatment for DVT, by comparing the DUS-detected recanalization rates and the occurrence of PTS. The secondary end-points of the analysis were the prevalence of pulmonary embolism, death, complications of treatment, and DVT relapse.

The statistical analyses were performed with SPSS 15.0 for Windows® (SPSS Inc., Chicago, IL), as percentages of patients and descriptive statistics. The χ2 test and Student's t test were used to compare univariate data and differences between groups. Linear and Cox's regressions were used in the univariate and multivariable analyses, and the results are reported as adjusted hazard ratios (HRs) with the accompanying 95% confidence intervals (CIs). ANOVA and a post hoc test were used in the analysis of groups. In all analyses, p values of < 0.05 were considered statistically significant.

ELIGIBILITY:
The noninclusion criteria were: pregnancy, age < 18 years or > 80 years, chronic renal failure, chronic hepatic chronic failure, inferior vena cava thrombosis, contraindication for any type of anticoagulation, previous DVT on the ipsilateral affected limb, or any type of active cancer, and patients who refused to participate in the study.

The exclusion criteria were: several hemorrhagic complications that required the discontinuation of anticoagulation, death after < 30 days, allergic reaction to any anticoagulant, a diagnosis of active cancer during follow-up, loss to follow-up, difficulty in achieving proper anticoagulation due to patient nonadherence to the treatment protocol, and incomplete data.

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
the long-term outcomes (after 12 months) in two groups of patients after treatment for DVT, by comparing the DUS-detected recanalization rates and the occurrence of PTS. | 6 months after the diagnosis of deep venous thrombosis.
  The patients are evaluated within 6 months with Duplex ultrasound to assess the recanalization rate. The criteria to assess Deep venous thrombosis are defined as as visualization of thrombus and/or lack of complete compressibility of the vein. Thrombus involving popliteal and/or more proximal veins was classified as proximal Deep venous thrombosis (DVT). The US findings in DVT include: the presence of echoes within the vascular lumen; the veins in axial scans are not compressible. Pulsed Doppler and duplex Doppler combine the morphologic and functional study. Injury caused by DVT at the valvular level (postphlebitic syndrome) is visualized. Venous segments were examined whether they were occluded, partially recanalized, or totally recanalized, and the development of venous reflux was evaluated.

SECONDARY OUTCOMES:
Clinical Signs and Symptoms in 84 patients.. | 6 months the diagnosis of deep venous thrombosis.
  The patients are evaluated within 6 months with clinical examination, to evaluate presence of pain in lower limbs, swelling and varicose veins. The post-thrombotic syndrome is characterized by aching pain on standing, dependent oedema, and the frequent develop-ment of brawny, tender induration of the subcutaneous tissues of the medial lower limb, a condition that has been termed lipodermatosclerosis. Pruritus and eczematous skin changes are frequently present, and a proportion of patients develop secondary superficial varicose veins as the syndrome evolves.Ulceration, often precipitated by minor trauma, arises in a considerable number of patients and is characteristically chronic and indolent with a high recurrence rate, once healing has been achieved. Uncommonly, patients with persistent obstruction may experience venous claudication, a bursting pain in the leg during exercise, which, in some respects,mimics arterial claudication (Immelman & Jeffrey, 1984).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Athayde Soares, MD, Dr/, Principal Investigator — Hospital do Servidor Publico Estadual
Locations (1):
- Hospital do Servidor Público Estadual de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We preserve confidential data.

REFERENCES:
- [Background] Rivaroxaban (Xarelto): Treatment of Venous Thromboembolic Events (Deep Vein Thrombosis [DVT], Pulmonary Embolism [PE]) and Prevention of Recurrent DVT and PE [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2015 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK344331/ PMID 26913324
- [Background] Isaacs AN, Doolin M, Morse C, Shiltz E, Nisly SA. Medication utilization evaluation of dabigatran and rivaroxaban within a large, multi-center health system. Am J Health Syst Pharm. 2016 Mar 1;73(5 Suppl 1):S35-41. doi: 10.2146/sp150031. PMID 26896524
- [Result] Finks SW, Trujillo TC, Dobesh PP. Management of Venous Thromboembolism: Recent Advances in Oral Anticoagulation Therapy. Ann Pharmacother. 2016 Jun;50(6):486-501. doi: 10.1177/1060028016632785. Epub 2016 Feb 25. PMID 26917821